CLINICAL TRIAL: NCT02407691
Title: Collaborative Care for the Detection and Management of Depression Among Adults Receiving Antiretroviral Therapy in South Africa: a Pragmatic Cluster Randomized Controlled Trial
Brief Title: Collaborative Care for the Detection and Management of Depression Among Adults Receiving Antiretroviral Therapy in South Africa
Acronym: COBALT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cape Town (Other)
Collaborators: King's College London (Other); University of KwaZulu (Other)
Responsible Party: Principal Investigator, Babalwa Zani, www.knowledgetranslation.co.za, University of Cape Town
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1R01MH100470-01 (NIH)
Record Dates: First submitted 2015-03-19; First posted 2015-04-03 (Estimated); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: HIV/AIDS; Depression; Chronic Diseases of Lifestyle
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Depression | interventions — Mental Health

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Primary Care 101 Enhanced guideline (Experimental): Primary Care 101 guideline with enhanced mental health
  Interventions: Other: Primary care 101 plus mental health
- Standard of care (Active Comparator): Primary Care 101 standard version guideline
  Interventions: Other: Standard Primary Care 101

INTERVENTIONS:
Other: Primary care 101 plus mental health — A facility-based stepped care intervention combining depression case detection by non-physician clinicians with group counselling intervention delivered by lay-health workers.
  Arms: Primary Care 101 Enhanced guideline
Other: Standard Primary Care 101 — Standard Primary Care 101 guideline with standard training
  Arms: Standard of care

SUMMARY:
With increasing access to antiretroviral therapy (ART) in South Africa, HIV has transitioned from a terminal illness to a long-term condition. It is likely to be accompanied by higher levels of disability and other chronic non-communicable diseases, resulting from the HIV itself, as well as adverse effects of medication. This requires an expansion of the purview of HIV care beyond direct HIV clinical care to also include a more comprehensive and integrated package of treatment and care for physical and mental conditions and their consequences. COBALT is a pragmatic cluster randomized controlled trial (RCT) in public sector primary care clinics in the North West Province of SA. It will assess mental health and HIV outcomes for depressed adults receiving ART by measuring the real-world effectiveness of a facility-based stepped care intervention combining depression case detection by non-physician clinicians with group counselling intervention delivered by lay-health workers.

ELIGIBILITY:
Inclusion Criteria:

Clinics:

1) 40 nurse-led primary care clinics providing ART in the Dr Kenneth Kaunda and Bojonala districts of the North West Province, South Africa

Patients:

1. Age ≥ 18 years and
2. Receiving ART at the time of enrollment and
3. Depressive symptoms, as indicated by a total score of 9 or more on the PHQ-9 and
4. Planning to reside in the area for the next year and
5. Capable of actively engaging in an interviewer-administered questionnaire at the time of recruitment, six and twelve months later and
6. Written consent to participate in the study

Exclusion Criteria:

Clinics:

1) Clinics which participate in the formative research and piloting of the intervention

Patients:

1) Inability to meet the above inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2002 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Viral load suppression | 12 months
  viral load value of <1000 RNA copies/ml
Patient Health Questionnaire 9 (PHQ-9) response | 6 months
  At least 50% improvement in PHQ-9 score compared with baseline

SECONDARY OUTCOMES:
PHQ-9 Response at 12 months | 12 months
  At least 50% improvement in PHQ-9 score compared with baseline
Depression Remission at 12 months | 12 months
  Score of less than 5 in PHQ-9
Mean PHQ-9 score at 6 and 12 months | 6 and 12 months
  Average score in the PHQ-9
Antiretroviral therapy programme retention | 12 months
  continuation in the ART programme
Viral load suppression at 12 months | 12 months
  Defined as a viral load of <400 copies/ml
Virological failure | 12 months
  Defined as two viral load values >1000 copies/ml
Appropriate maintenance on enrollment ART regimen OR ART regimen switched to second-line | 12 months
  continuation with the ART regimen OR change
ART adherence | 12 months
  30 day VAS self reported measure
Change in viral load values over time | 12 months
  change in HIV RNA copies measured by PCR
Depression severity (categorised as mild, moderate, moderately severe or severe depression at 6 and 12 months) | 6 and 12 months
  Mild depression defined as a score of 5 to 9; moderate depression defined as a score of 10-14 Moderately severe depression defines as a core of 15-19, and Severe depression defined as a score of 20-27.
Antidepressant treatment initiated or intensified | 12 months
  start or intensification of anti-depressants after baseline
Counselling for depression by a clinic-based counsellor | 12 months
  Having counselling sessions with the clinic counsellor
Referral to specialist mental health worker/service | 12 months
  Referral by a nurse to mental health worker/service
Hospital admissions | 12 months
  number and duration of overnight hospital stays
Mortality | 12 months
  Mortality reported at loss to follow-up or through the South African Population register
Stress | 12 months
  Measured through the Percieved Stress Scale
Stigma | 12 months
  Measured through the 6-item AIDS related stigma scale
Risk factors for cardiovascular diseases | 12 months
  Measured by blood pressure, weight, smoking status
Detection and treatment of other chronic diseases | 12 months
  Identification of new cases of NCDs or risk factors of Chronic deseases
Provision of integrated care from patient perspective | 12 months
  Assessed using the Patient Assessment of Care for Chronic Conditions (PACIC)

OTHER OUTCOMES:
Disability | 12 months
  Measured by WHODAS 2
Care utilization and resource use | 12 months
  Measured by service use questionnaire
Productivity and economic measures | 12 months
  Self reported

CONTACTS AND LOCATIONS:
Overall Officials: Lara Fairall, PhD, Principal Investigator — University of Cape Town, Cape Town, South Africa; Inge Pitersen, PhD, Principal Investigator — University of KwaZulu-Natal, Durban, South Africa; Graham Thornicroft, PhD, Principal Investigator — King's College London
Locations (2):
- South Africa (2):
  - Dr Kenneth Kaunda District, Klerksdorp, North West
  - Bojanala District, Rustenburg, North West

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zani B, Fairall L, Petersen I, Folb N, Bhana A, Thornicroft G, Hanass-Hancock J, Selohilwe O, Petrus R, Carmona S, Lombard C, Lund C, Levitt N, Bachmann M. Sociodemographic and health-related factors associated with viral load non-suppression and body mass index in adults with depression symptoms receiving antiretroviral therapy in South African primary care: secondary analysis of randomised trial data. medRxiv [Preprint]. 2025 Aug 5:2025.08.01.25332690. doi: 10.1101/2025.08.01.25332690. PMID 40799963
- [Derived] Zani B, Fairall L, Petersen I, Folb N, Bhana A, Hanass-Hancock J, Selohilwe O, Petrus R, Georgeu-Pepper D, Mntambo N, Kathree T, Carmona S, Lombard C, Lund C, Levitt N, Bachmann M, Thornicroft G. Effectiveness of a task-sharing collaborative care model for the detection and management of depression among adults receiving antiretroviral therapy in primary care facilities in South Africa: A pragmatic cluster randomised controlled trial. J Affect Disord. 2025 Feb 1;370:499-510. doi: 10.1016/j.jad.2024.10.061. Epub 2024 Oct 21. PMID 39442695
- [Derived] Fairall L, Petersen I, Zani B, Folb N, Georgeu-Pepper D, Selohilwe O, Petrus R, Mntambo N, Bhana A, Lombard C, Bachmann M, Lund C, Hanass-Hancock J, Chisholm D, McCrone P, Carmona S, Gaziano T, Levitt N, Kathree T, Thornicroft G; CobALT research team. Collaborative care for the detection and management of depression among adults receiving antiretroviral therapy in South Africa: study protocol for the CobALT randomised controlled trial. Trials. 2018 Mar 22;19(1):193. doi: 10.1186/s13063-018-2517-7. PMID 29566739
- See also: Related Info — http://www.knowledgetranslation.co.za